CLINICAL TRIAL: NCT05866419
Title: Safety and Performance of the ThecaFlex DRx™ System Port and Catheter for Chronic Intrathecal Access, Cerebrospinal Fluid (CSF) Aspiration, and DElivery of Nusinersen in Spinal Muscular Atrophy (SMA) Patients Resistant to Lumbar PunctuRE Trial (PIERRE)
Brief Title: Study of an Intrathecal Port and Catheter System for Subjects With Spinal Muscular Atrophy
Acronym: PIERRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcyone Therapeutics, Inc (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT-0179
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Spinal Muscular Atrophy; Spine Deformity; Scoliosis
MeSH Terms: conditions — Muscular Atrophy, Spinal; Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ThecaFlex DRx Port and Catheter System (Experimental): Subjects who meet all of the inclusion and none of the exclusion would be eligible to receive the ThecaFlex DRx Port and Catheter System.
  Interventions: Device: ThecaFlex DRx System

INTERVENTIONS:
Device: ThecaFlex DRx System — The ThecaFlex DRx™ System consists of an implantable intrathecal catheter, and an implantable subcutaneous port, designed specifically to meet the implantation, Cerebrospinal Fluid (CSF) aspiration, and intrathecal delivery and dosing needs of patients (aged ≥ 3 years) requiring repeated/on-going intermittent chronic bolus intrathecal treatment for life threatening, debilitating Central Nervous System (CNS) disorders who are precluded from Lumbar Puncture (LP) due to complex spine conditions, or who are resistant to LP for therapy administration or CSF aspiration.

SUMMARY:
The primary objective of the clinical investigation is to demonstrate successful clinical use of the ThecaFlex DRx™ System in delivering nusinersen in subjects with spinal muscular atrophy (SMA).

All enrolled subjects will undergo implantation of the investigational device (ThecaFlex DRx™ System) and will be followed for 12 months after receiving the implant. The 12-month data will be used to assess the primary endpoint support a Pre-Market Approval (PMA) application.

DETAILED DESCRIPTION:
This is a multicenter, multi-national, prospective, non-randomized, single arm, group sequential design, pivotal clinical investigation (device exemption study) to assess the safety and performance of the ThecaFlex DRx™ System in subjects with SMA.

The subject population will include subjects aged ≥ 3 years with SMA who are considered candidates for intrathecal port and catheter implantation because they require chronic, bolus intrathecal administration of necessary therapy, and who meet all the inclusion/exclusion criteria for the clinical investigation.

After a screening period of up to 200 days, all enrolled subjects will undergo implantation of the investigational device (ThecaFlex DRx™ System) and will be followed for 12 months after receiving the implant.

In agreement with the nusinersen dosing information, the treatment frequency will be adapted for non-naïve and naïve subjects:

Subjects who are not naïve to nusinersen should have nusinersen maintenance doses administered via the implant every 4 months (i.e., 4, 8, and 12 months after their last nusinersen dose, before enrollment in the clinical investigation).

Subjects who are naïve to nusinersen will have their first three loading doses administered via the implant at 14-day intervals. The fourth loading dose should be administered 30 days after the third dose. A maintenance dose should be administered once every 4 months thereafter within the 12 months post-implantation.

A DMC and Clinical Events Committee (CEC), independent of each other and the Sponsor, will be used to perform ongoing consistent adjudication of events related to the safety throughout the entire duration of the clinical investigation and to periodically review data that relate to the safety of the study.

The clinical investigation will enroll 90 subjects. The clinical investigation incorporates a lead-in phase which consists of 10 subjects enrolled, implanted, and followed for 30-days. Enrollment for the lead-in phase is expected to take approximately 6 to 9 months, at which point the Data Monitoring Committee (DMC) will review the data for safety and approve continuation of enrollment. The second phase of enrollment is expected to take approximately 12 to 15 months.

Individual subjects are anticipated to be enrolled in the clinical investigation for approximately 37 months. The total duration of this clinical investigation is estimated to be approximately 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 3 years or older
2. Subject diagnosed with SMA who are candidates for Spinraza treatment as indicated in its label
3. Subject resistant to lumbar puncture (LP), where resistance is defined as:

   1. Subject with respiratory issues or other comorbidities who is at an increased risk for complications due to the need for repeat anesthesia and imaging radiation exposure to safely perform LP; or
   2. Subjects for whom the treating physician determines implantation of the ThecaFlex DRx™ System is otherwise in the subject's best interest
4. Subject has been prescribed nusinersen via chronic intrathecal bolus administration in accordance with the drug labeling and first port access of the ThecaFlex DRx system is planned within 2 weeks of implantation
5. Subject, per Investigator discretion, is able to undergo a percutaneous or open surgical procedure for index port and catheter implantation where at least 7 cm of the ThecaFlex DRx system catheter will be placed intrathecally
6. Subject (or subject's legally authorized representative) is willing and able to provide written informed consent; and
7. Subject and parent/caregiver able and willing to complete all clinical investigation procedures, measurements, and visits.

Exclusion Criteria:

1. Subject meets any of the contraindications for use of the ThecaFlex DRx™ System as outlined in the ThecaFlex DRx™ System Instructions for Use
2. Presence or history of (< 6 months prior to the procedure): an implanted microinfusion pump, intrathecal catheter, or other intrathecal drug delivery devices/component, or implanted shunt for drainage of cerebrospinal fluid (CSF), or reservoir in the CSF space (note: any ThecaFlex Port and Catheter System must not be placed in the same location as a previous indwelling port and catheter)
3. Subject is pregnant or nursing or plans to become pregnant during the course of the clinical investigation
4. Any condition or event, which in the opinion of the Investigator may adversely affect the safety and effective implantation and use of the ThecaFlex DRx™ system or confound the clinical investigation, including:

   1. Severe structural impediment that may preclude safe implantation of the catheter and port
   2. Major medical events within 60 days prior to screening; or
   3. Relevant surgeries (e.g., head and neck, back, etc.) within 60 days prior to screening or planned during the duration of the clinical investigation
   4. Space-occupying lesion with mass effect
   5. Posterior fossa mass
   6. Arnold-Chiari malformation
   7. Coagulation abnormalities and/or thrombocytopenia
   8. Insufficient or inadequate skin or underlying fat to adequately protect the port or enough surface area to allow the skin to close safely
5. Subject is contraindicated for administration of nusinersen per its approved labeling
6. History of intrathecal granuloma formation
7. History of bacterial meningitis or aseptic meningitis within 6 months of screening
8. History of tumors or other spinal abnormalities documented by magnetic resonance imaging (MRI) or computed tomography (CT) that would interfere with the catheter implantation procedures or CSF circulation
9. History of hydrocephalus
10. Diagnosed degenerative muscular disease other than SMA
11. History of depression, cognitive impairment, or another psycho-behavioral problem that in the opinion of the Investigator may preclude safe participation in the clinical investigation and
12. Serious medical condition that, in the opinion of the investigator, may lead to reduced life expectancy beyond 12 months.
13. Subject is involved in another Investigation Device Exemption Study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with successful Implantation of the ThecaFlex DRx™ Port and Catheter | 12 Months
  The primary outcome measures the proportion of subjects with successful implantation of the ThecaFlex DRx™ Port and Catheter System who are able to receive successful intrathecal therapy infusion(s).
The proportion of subjects with successful Intrathecal Therapy Infusion(s) through 12 months | 12 Months

SECONDARY OUTCOMES:
Proportion of subjects with reduced anesthesia and radiation exposure compared to repeat LP for nusinersen infusion in SMA subjects. | 12 months
Incidence of device-related adverse events (AEs)/complications through 12 months | 12 months
Incidence of procedural complications through 12 months | 12 months
Incidence of nusinersen-related AEs | 12 months
Mean duration of radiation exposure from implant through 12-month follow-up | 12 months

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Children's Hospital Orange County, Orange, California
  - Stanford Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Lurie Childrens Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Columbia University Irving Medical Center/NewYork Presbyterian Hospital, New York, New York
  - UH Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Childrens Hospital of the King's Daughters, Norfolk, Virginia
- Universitätsklinikum Essen, Essen, Germany
- Centro Clinico Nemo, Milan, Italy
- Poland (2):
  - Specialised Hospital Ludwika Rydygiera, Krakow
  - Research Institute of Polish Mother's Memorial Hospital, Lodz
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politecnico la Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No